CLINICAL TRIAL: NCT01360905
Title: Study to Determine the Equivalence of the Monica AN24 Monitor to Predicate Devices for (FHR) and (UC) During Pre-term Labor and Multiples
Brief Title: Study to Support Fetal Heart Rate and Uterine Contraction for Preterm Labor in Singleton and Multiple Pregnancies
Status: Terminated | Type: Observational
Why Stopped: Difficulty in recruiting
Sponsor: Monica Healthcare Ltd (Industry)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 100_CT-045
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Pre Term Labor; Multiple Pregnancy
Keywords: PTL; Multiples

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the Monica AN24 fetal monitor to previously FDA approved devices for Fetal Heart Rate and Uterine Contractions in labor for Multiples and pre term labor.

DETAILED DESCRIPTION:
Clinical Investigation for a non-inferiority/equivalence study that aims to determine the acceptable performance of the Monica AN24 during the first and when possible the second stages of labor by determining whether the Monica AN24 fetal heart rate (FHR) and uterine contractions (UC) monitoring device is non-inferior/equivalent to Doppler FHR and tocodynamometer UC using direct fetal scalp electrode (FSE) FHR and intrauterine pressure catheter (IUPC) UC as a reference, either collected simultaneously with the Monica and Doppler FHR/tocodynamometer UC data, or from previous studies to define the expected accuracy and success rate when comparing Monica FHR and UC with Doppler FHR and tocodynamometer UC respectively

ELIGIBILITY:
Inclusion Criteria:

* She is >=24weeks 0days but less than 36 completed weeks, with a singleton pregnancy or >=34weeks 0days with a multiple pregnancy and has been admitted to the Labor and Delivery Unit
* She is in the latent phase of spontaneous labor, or has been admitted for induction of labor
* She has given her informed consent to participate as a subject
* She has none of the exclusion criteria

Exclusion Criteria:

* Known major fetal malformation or chromosome abnormality
* Involvement in another clinical trial currently or previously in this pregnancy
* Medical or obstetric problem that would preclude the use of abdominal electrodes (e.g., skin eruptions, sensitivity to adhesives)
* Significant medical or obstetric problem that in the investigator's opinion would make the woman incapable of taking part in the study

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is women of >= 24 weeks of singleton pregnancy or women of >=24 weeks of multiple pregnancy, that have been admitted to the Labor and delivery suite
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
equivalence with predicate device | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Mizra, Dr, Principal Investigator — New York Presbytarian Hospital
Locations (1):
- Columbia University Medical Center, New York, New York, United States